CLINICAL TRIAL: NCT05364619
Title: Qingre Huashi Granules Combined the Modified Dual Therapy for Helicobacter Pylori Infection Treatment in the Elderly Patient, a Multi-center, Randomized, Controlled Trial
Brief Title: Qingre Huashi Granules Combined the Modified Dual Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University International Hospital (Other); Beijing Geriatric Hospital (Other); Beijing Changping Integrative Medicine Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShouFa-2022-2-40711
Record Dates: First submitted 2022-04-24; First posted 2022-05-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Geriatic; Dual therapy; Bismuth-containing quadruple therapy; Qingre Huashi Decoction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QHD group (Experimental): Qingre Huashi Granules 1 package twice daily, Rabeprazole 20mg triple daily, Amoxycillin 1g triple daily. The duration is 14 days.
  Interventions: Drug: Qingre Huashi Granules combined the modified dual therapy
- Control group (Active Comparator): Rabeprazole 20mg twice daily, bismuth potassium citrate 220mg twice daily, Amoxycillin 1g twice daily, clarithromycin 500mg twice daily. The duration is 14 days.
  Interventions: Drug: Bismuth containing quadruple therapy

INTERVENTIONS:
Drug: Qingre Huashi Granules combined the modified dual therapy — Qingre Huashi Granules combined the modified dual therapy for 14 days
  Arms: QHD group
Drug: Bismuth containing quadruple therapy — Bismuth containing quadruple therapy for 14 days
  Arms: Control group

SUMMARY:
This is an open-label, randomized controlled trial. The aim of the study is to evaluate the efficacy and safety of the Qingre Huashi Granules combined the modified dual therapy (or called high dose dual therapy) for Helicobacter pylori infection specifically in geriatric patients, compared with the bismuth containing quadruple therapy. A total of 160 eligible patients will be enrolled in 4 hospitals. The eradication rate, symptoms, and the adverse events will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Current Helicobacter pylori infection.
* Age ≥ 60 years.
* Diagnosed with syndrome of dampness-heat by Traditional Chinese Medicine.
* Signed the informed consent document.

Exclusion Criteria:

* History of Helicobacter pylori treatment.
* History of gastric surgery.
* Allergic to any medications involved in the intervention.
* Sever complications, such as lung dysfunction, uncontrolled hypertension, diabetes, cardiovascular disease, renal dysfunction (eGFR<60ml/min'1.73m2) , malignant tumor，mental disorder.
* Taking medications that may be conflict to the intervention drugs.
* Failing to express symptoms, unwilling to cooperate.
* Taking any antibiotics within a month.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | The 4th week after the treatment.
  At the 4th week after the treatment, the 13-carbon urease test was conducted to evaluate the eradication condition. The value of "delta over baseline" <4 was considered to be successful eradication.

SECONDARY OUTCOMES:
7-point Global Overall Symptom Scale | Baseline, the second and sixth week after the treatment, respectively.
  The 7-point Global Overall Symptom Scale was used to record and evaluate the symptoms. The scale value ranges from 7 to 56. The higher scale means the worse outcome.
Efficacy Scale of the Dampness-heat syndrome | Baseline, the second and sixth week after the treatment, respectively.
  The Scale of the Dampness-heat syndrome was used to record and evaluate the symptoms related to the Traditional Chinese Medicine symptoms. The scale value ranges from 0 to 24. The higher scale means the worse outcome.
Adverse events rate | During the follow-up, up to 6 weeks.
  Any adverse event related to the drugs will be recorded during the entire follow-up period.

OTHER OUTCOMES:
CYP2C19 Genotype | The sixth week after the treatment.
  Failed cases will receive the CYP2C19 Genotype test.
Helicobacter pylori antibody test. | Baseline
  The antibody of anti-UREA, anti-UREB, anti-CagA, and anti-VacA was tested.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Changping Integrative Medicine Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided